CLINICAL TRIAL: NCT06699420
Title: The Efficacy and Safety of Qishenyiqi Dripping Pill in Patients With Coronary Microvascular Disease
Brief Title: Qishenyiqi Dripping Pill for Coronary Microvascular Disease
Acronym: CMVD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Prof., Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qishenyiqi for CMVD
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qishenyiqi Dripping Pill (Experimental)
  Interventions: Drug: Qishenyiqi dripping pills 1 bag, three times a day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo 1 bag, three times a day

INTERVENTIONS:
Drug: Qishenyiqi dripping pills 1 bag, three times a day — Qishenyiqi dripping pills, 1 bag once, three times a day, 12 months
  Arms: Qishenyiqi Dripping Pill
Drug: Placebo 1 bag, three times a day — Placebo, 1 bag once, three times a day, 12 months
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of Qishenyiqi in patients with microvascular angina pectoris. Long-term follow-up of 1 year will be performed to evaluate the effect of Qishenyiqi on coronary flow reserve and adverse cardiovascular events in patients with coronary microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Repeated chest pain attacks with typical exertional angina pectoris or resting angina pectoris attacks;
* Coronary normal or stenosis < 20%;
* Ischemic depression in ST segment during resting or exercise;
* Blood flow reserve (CFR) of the anterior descending coronary artery < 2.0;
* Subjects or their guardians agreed to participate in this study.

Exclusion Criteria:

* Previous myocardial infarction or PCI or CABG treatment;
* A history of heart failure;
* Severe arrhythmia;
* Refractory hypertension or hypertension accompanied by left ventricular wall thickness > 12 mm;
* Familial hypercholesterolemia;
* Takayasu arteritis, Kawasaki disease or coronary artery malformation;
* Pregnant or nursing, or having the intention to give birth within one year;
* Hepatic or renal dysfunction;
* Allergic to contrast agents or traditional Chinese medicines;
* Patients who participated in clinical research of other drugs within 3 months before being selected.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of coronary flow reserve measured by three-dimensional echocardiography from baseline to 12 months after follow-up | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Qianfoshan Hospital, Shandong University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No